CLINICAL TRIAL: NCT06620783
Title: The Efficacy of an Exercise Program and a Yoga Program in Mitigating Stress and Improving Mental Health Among Employees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Boramae Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-2309-855-301
Record Dates: First submitted 2023-10-19; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2023-10

CONDITIONS: Depression; PTSD; Work Related Stress
MeSH Terms: conditions — Depression; Stress Disorders, Post-Traumatic; Occupational Stress | interventions — Exercise; Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- exercise program group (Active Comparator): Those in the exercise program group will access and undertake the exercise program on a web or mobile platform for approximately 50 minutes per session, three times a week, for a total of 12 sessions over 4 weeks.
  Interventions: Behavioral: exercise
- yoga program group (Active Comparator): The yoga program group will access and perform the yoga program on a web or mobile platform for approximately 50 minutes per session, three times a week, for a total of 12 sessions over 4 weeks.
  Interventions: Behavioral: yoga
- self-care group (Sham Comparator): The self-care group will access materials helpful for stress management via a web or mobile platform and engage in self-study three times a week, for a total of 12 sessions over 4 weeks.
  Interventions: Behavioral: active self-care

INTERVENTIONS:
Behavioral: exercise — Those in the exercise program group will access and undertake the exercise program on a web or mobile platform for approximately 50 minutes per session, three times a week, for a total of 12 sessions over 4 weeks.
  Arms: exercise program group
Behavioral: yoga — The yoga program group will access and perform the yoga program on a web or mobile platform for approximately 50 minutes per session, three times a week, for a total of 12 sessions over 4 weeks.
  Arms: yoga program group
Behavioral: active self-care — The self-care group will access materials helpful for stress management via a web or mobile platform and engage in self-study three times a week, for a total of 12 sessions over 4 weeks.
  Arms: self-care group

SUMMARY:
To reduce workplace stress and promote mental health, participants were divided into three groups: exercise program, yoga program, and self-care. The effectiveness of the exercise and yoga programs was evaluated using pre- and post-program self-reported questionnaires, HRV (Heart Rate Variability), and 2-lead EEG.

DETAILED DESCRIPTION:
After screening, a preliminary assessment is conducted on the study participants who have agreed to participate. The preliminary assessment includes medical history review, questionnaires related to current physical activity levels, mental health-related questionnaires concerning stress, depression, insomnia, job stress, and job burnout. It also includes tests for heart rate variability (HRV), physiological stress-related indicators via a 2-lead EEG, and a basic physical ability assessment. After the preliminary evaluation:

Those in the exercise program group will access and undertake the exercise program on a web or mobile platform for approximately 50 minutes per session, three times a week, for a total of 12 sessions over 4 weeks.

The yoga program group will access and perform the yoga program on a web or mobile platform for approximately 50 minutes per session, three times a week, for a total of 12 sessions over 4 weeks.

The self-care group will access materials helpful for stress management via a web or mobile platform and engage in self-study three times a week, for a total of 12 sessions over 4 weeks.

After completing their respective programs, participants from the exercise group, yoga group, and the self-care control group will revisit the hospital within a week to undergo the same tests as in the preliminary evaluation, excluding medical history and physical activity information. Moreover, to determine whether the effects of the exercise and yoga programs persist after the program ends, participants will return for the same tests one month after the 4-week program concludes. Using the data obtained, the study will measure the changes induced by the self-directed exercise and yoga programs on the participants' clinical scales like stress, symptoms of depression, HRV, EEG, and basic physical abilities. The effects on the improvement of psychological and physiological stress indicators of the self-care group, using stress data, will then be compared and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Employed individuals aged 19 to 49 years.
* Participants with moderate stress levels, scoring 14 or higher on the Perceived Stress Scale.
* Individuals currently undergoing pharmacological treatment for psychiatric conditions such as depression, anxiety disorders, or insomnia, provided they are in a stable phase with no expected changes in medication dosage during the clinical trial period.
* Participants who fully understand the clinical trial protocol and have voluntarily consented to participate.

Exclusion Criteria:

* Adults under the age of 19 or over the age of 49.
* Individuals with dementia, intellectual disabilities, or other cognitive impairments.
* Those with neurological disorders such as epileptic conditions, stroke, or other neurological diseases.
* Individuals with a history of, or currently diagnosed with, psychiatric disorders like schizophrenia or bipolar disorder.
* Individuals with a history of suicidal ideation or attempts.
* Those taking medications or having conditions determined by the research team to potentially affect the reliability of the HRV (Heart Rate Variability) test (e.g., heart disease, pulmonary disease, etc.).
* Those who have received non-pharmacological psychiatric treatment or counseling in the current or past 6 months.
* Individuals deemed by the research team to have physical limitations that make it difficult to participate in exercise or yoga programs.

Ages: 19 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2023-10-04 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Stress level | Pre-intervention, Post-intervention (right after the 4 weeks of intervention, within at most a week timeframe), 1 month follow-up
  Stress level by the Perceived Stress Scale. We will use the Korean version of the Perceived Stress Scale, originally developed by Cohen et al. (1983) and revised by Cohen et al. in 1988. This version has been adapted into Korean and validated to measure participants' perceived stress experiences. The total score ranges from 0 to 40, with each item rated on a 5-point Likert scale from 0 (never) to 4 (very often). A higher score indicates a greater perception of unpredictability, lack of control, and overwhelming stress-related experiences over the past month.
Depression level | Pre-intervention, Post-intervention (right after the 4 weeks of intervention, within at most a week timeframe), 1 month follow-up
  Depression level by the Patient Health Questionnaire 9. This is a self-report assessment tool designed to briefly screen for depressive disorders and evaluate the severity of depressive symptoms (Kroenke et al., 2001). It comprises items corresponding to the nine diagnostic criteria for major depressive disorder according to the DSM-IV, based on depressive symptoms experienced over the past two weeks. The total score ranges from 0 to 27, with higher scores indicating more severe depressive symptoms. Scores of 5 or above, 10 or above, 15 or above, and 20 or above suggest mild, moderate, moderately severe, and severe depression, respectively.

SECONDARY OUTCOMES:
Insomnia level | Pre-intervention, Post-intervention (right after the 4 weeks of intervention, within at most a week timeframe), 1 month follow-up
  Insomnia level by the Insomnia severity index. This self-report scale, developed by Morin (1993), assesses the severity of insomnia based on the diagnostic criteria of the DSM-IV and the International Classification of Sleep Disorders (ICSD). It consists of seven items evaluating the type and severity of insomnia over the past two weeks, including sleep satisfaction, daytime functioning impairment, sleep-related difficulties, and distress caused by sleep problems. The total score ranges from 0 to 28, with scores of 8 to 14 indicating mild insomnia, 15 to 21 indicating moderate clinical insomnia, and 22 or above indicating severe insomnia.
PTSD symptoms | Pre-intervention, Post-intervention (right after the 4 weeks of intervention, within at most a week timeframe), 1 month follow-up
  To measure the level of PTSD symptoms in study participants, we will use the PTSD Checklist for DSM-5 (PCL-5), developed by Weathers et al. (2013), based on the diagnostic criteria of the DSM-5. The PCL-5 is an adaptation of the PTSD Checklist (PCL), originally created by Weathers et al. (1993), and was translated by Park et al. (2016) and validated by Lee et al. (2020). The PCL-5 assesses the severity of symptoms experienced over the past month due to a past traumatic event. It consists of 20 items rated on a 5-point Likert scale (0 = Not at all, 4 = Extremely), with higher scores indicating more severe PTSD symptoms. The PCL-5 includes subscales for intrusion, avoidance, negative alterations in cognition and mood, and hyperarousal. The provisional cutoff score is known to be between 31 and 33, with a cutoff of 25.5 identified in a validation study of the general Korean adult population (Lee et al., 2022; Bovin et al., 2016).
Work-related stress levels | Pre-intervention, Post-intervention (right after the 4 weeks of intervention, within at most a week timeframe), 1 month follow-up
  This tool is the shortened version of the Korean Occupational Stress Scale (KOSS), originally consisting of 43 items, now reduced to 24 items. Each item is rated on a 5-point Likert scale ranging from 1 (Not at all) to 5 (Very much). Higher scores indicate higher levels of job stress experienced over the past month. The scale covers seven domains: job demands, job autonomy, job insecurity, interpersonal conflict, organizational system, inadequate compensation, and workplace culture. It was designed for easy application in field settings (Jang Se-jin et al., 2005).
Burnout symptoms | Pre-intervention, Post-intervention (right after the 4 weeks of intervention, within at most a week timeframe), 1 month follow-up
  To measure the current level of job burnout in the study participants, we will use the Maslach Burnout Inventory-General Survey (MBI-GS), developed by Schaufeli et al. (1996) to assess burnout in general workers, and adapted and validated by Shin Kang-hyun (2003). This scale evaluates the three core dimensions of burnout syndrome experienced in the workplace: exhaustion, cynicism, and professional efficacy. Each dimension consists of five items, rated on a 7-point Likert scale from 0 (strongly disagree) to 6 (strongly agree). Higher scores in the exhaustion and cynicism dimensions, and lower scores in the professional efficacy dimension, indicate greater levels of job burnout.
Emotional states | Pre-intervention, Post-intervention (right after the 4 weeks of intervention, within at most a week timeframe), 1 month follow-up
  To measure participants' positive and negative affect, we will use the revised Korean version of the Positive and Negative Affect Schedule (K-PANAS-R). This scale was originally developed by Watson et al. (1988) and was validated in Korean by Lee Hyun-hee et al. (2003). Park Hong-seok et al. (2016) reviewed its limitations and revised the scale through translation and back-translation of the original. The K-PANAS-R assesses emotions experienced by participants over the past week using 20 items, each rated on a 5-point Likert scale, reflecting the intensity of the emotions described by the adjectives.
Basic physical level | Pre-intervention, Post-intervention (right after the 4 weeks of intervention, within at most a week timeframe), 1 month follow-up
  To assess baseline physical fitness levels, the following tests, as recommended by the Korean Society of Sports Science, were conducted and the respective results were recorded: flexibility, muscle strength, knee push-up, gait test, and balance test.
2-lead EEG | Pre-intervention, Post-intervention (right after the 4 weeks of intervention, within at most a week timeframe), 1 month follow-up
  For measuring neural activity in the prefrontal lobe, we will use a 2-channel EEG (FP1, FP2). EEG is a non-invasive method that quantifies brain electrical activity by attaching electrodes to the scalp to capture electrical signals generated by potential differences. This method is non-invasive, offers excellent temporal resolution, and is cost-effective, making it widely applicable in studies involving general populations. The raw data collected by the device are processed using TeleScan (© Laxtha, Inc.) to calculate absolute power, frequency ratio, relative power, and symmetry across different frequency bands. The key indicators derived from the data include: Theta, Alpha, Low-Beta, Mid-Beta, High-Beta, Gamma, the (Low-Beta + Mid-Beta)/Theta power ratio, and the Alpha/High-Beta power ratio.
Heart rate variability | Pre-intervention, Post-intervention (right after the 4 weeks of intervention, within at most a week timeframe), 1 month follow-up
  Heart rate variability (HRV) is an effective method for quantitatively assessing autonomic nervous system activity and balance. It is widely used to examine changes in autonomic activity and balance caused by stress, as well as to gather information on stress-related disorders. HRV can be analyzed using various methods, with time domain analysis and frequency domain analysis being the most commonly employed. In this study, we will use several frequently used indicators from frequency domain analysis in HRV research, including: TP (total power), LF (low frequency), HF (high frequency), and the LF/HF+LF ratio.

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul Metropolitan Government-Seoul National University Boramae Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No